CLINICAL TRIAL: NCT06002230
Title: Use of Homeopathy in Patients Suffering From Long COVID-19 (LONGCOVIHOM): A Retrospective Case Series
Brief Title: Use of Homeopathy in Patients Suffering From Long COVID-19
Acronym: LONGCOVIHOM
Status: Completed | Type: Observational
Sponsor: Michael Frass (Other)
Collaborators: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor-Investigator, Michael Frass, Clinical professor, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 111
Record Dates: First submitted 2023-08-18; First posted 2023-08-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Adjustment Reaction With Physical Symptoms
Keywords: Complementary therapy; Homeopathy; COVID-19; Long-COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Homeopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with individualized homeopathy: Patients suffering from symptoms of Long COVID-19 were treated with individualized homeopathy.
  Interventions: Drug: Homeopathic medicines

INTERVENTIONS:
Drug: Homeopathic medicines — Globules were administered orally..
  Other Names: Homeopathic medicinal products

SUMMARY:
In some patients, coronavirus (COVID-19) can cause symptoms that last weeks or even months after the infection has gone. The aim of this study was to describe the effect of adjunctive individualized homeopathic treatment delivered to Long-COVID-19 patients with previously confirmed symptomatic SARS-CoV-2 infection.

DETAILED DESCRIPTION:
All patients had been tested positive for SARS-CoV-2 before having developed Long-COVID-19 symptoms. Several testing methods were carried out in each patient to analyze a SARS-CoV-2 infection. For a confirmed infection, at least 3 out of these 5 tests had to be positive. Tests for the orthomyxoviruses influenza A and B, human metapneumovirus (hMPV) and paramyxoviruses were negative unless stated otherwise.

The homeopathic physician treated all Long-COVID-19 patients by individualized homeopathy. Repertorization of the symptoms of the current pandemic and a search in the current homeopathic literature on COVID-19 was performed using computer program. All available homeopathic medicinal products (HMPs) could be chosen by the treating physician.

Modified MONARCH criteria were assessed post hoc by all authors. Deviations were solved by discussion in person. Clinical outcome of case reports was evaluated using the "Modified Naranjo Criteria for Homeopathy-Causal Attribution Inventory". Eight points is assumed as the limit for potential correlation between homeopathic therapy and amelioration of the symptoms or healing in chronic cases.

ELIGIBILITY:
Inclusion Criteria:

Long COVID-19 symptoms following recovery from SARS-CoV-2 infection

Exclusion Criteria:

Patients not signing informed consent

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Long COVID-19 symptoms following recovery from SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Modified Naranjo criteria | 3 days
  10 Naranjo criteria are evaluated, eight points is assumed as the limit for potential correlation between homeopathic therapy and amelioration of the symptoms or healing in chronic cases.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, MD, Study Director — Institute for Homeopathic Research
Locations (1):
- Sigmund Freud Private University, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided